CLINICAL TRIAL: NCT04480242
Title: Assessment of Children and Adolescents With Asthma: An Observational Prospective Study
Brief Title: Asthma Research in Children and Adolescents
Acronym: ARCA
Status: Active, not recruiting | Type: Observational
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Sponsor
Other Study IDs: ARCA2017; PI15/00449 (Other Grant/Funding Number: Instituto Salud Carlos III Fondo Europeo Desarrollo Regional)
Record Dates: First submitted 2020-07-13; First posted 2020-07-21 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-05

CONDITIONS: Persistent Asthma; Asthma in Children; Asthma Exacerbation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Asthma Research in Children and Adolescents - Spanish Cohort: Groups defined according to treatments prescribed during regular clinical practice and to the exposure to inhalation techniques monitoring
  Interventions: Drug: Inhaled Corticosteroids (ICs); Drug: Fixed-Dose Combination of Inhaled Corticosteroids and Long- Acting Beta-agonist (ICs/LABA); Drug: Other treatments; Drug: Inhaler device; Behavioral: Regularly monitoring of the Inhalation technique through mobile app

INTERVENTIONS:
Drug: Inhaled Corticosteroids (ICs) — Any corticosteroid (beclomethasone, budesonide, ciclesonide, fluticasone propionate, fluticasone furoate, mometasone, and triamcinolone) prescribed by the pediatrician as an inhaled controller medication, for daily management of asthma. The daily dose of ICs prescribed will be translated into beclomethasone equivalent.
  Other Names: Treatments prescribed during regular clinical practice
Drug: Fixed-Dose Combination of Inhaled Corticosteroids and Long- Acting Beta-agonist (ICs/LABA) — Beclomethasone/formoterol, budesonide/formoterol, fluticasone furoate/vilanterol, fluticasone propionate/formoterol, fluticasone propionate/salmeterol, and mometasone/formoterol. Any of these combinations prescribed by the pediatrician as an inhaled controller medication, for daily management of asthma.
  Other Names: Treatments prescribed during regular clinical practice
Drug: Other treatments — Low-dose oral corticosteroids, long-acting muscarinic antagonist (tiotropium), low-dose macrolides (azithromycin), leukotrienes receptor antagonists (i.e. montelukast), or biologic agents (i.e. omalizumab).
  Other Names: Treatments prescribed during regular clinical practice
Drug: Inhaler device — Pressurized metered-dose inhalers (pMDIs), Breath-actuated pMDIs, Dry powder inhalers (DPIs), Nebulizers, Soft Mist Inhalers.
  Other Names: Treatments prescribed during regular clinical practice
Behavioral: Regularly monitoring of the Inhalation technique through mobile app — App users are randomized within each pediatrician into two groups of equal size defined within the subsample recruited, so that 50% of the participants are allocated to answer the inhalation techniques, and the other 50% are allocated to answer the environment support scales. Once the app is downloaded, at month 2 and every 6 months thereafter the intervention group answers the inhalation techniques scale (group 1) and the control group answers the environment support scale (group 2).

SUMMARY:
The purpose of this study is to assess the evolution of disease control, health-related quality of life, and the risk of severe asthma exacerbations in children and adolescents with persistent asthma in Spain at short, mid and long-term follow-up. Patient-reported information in this project is collected by computer assisted telephone interviews (CATI) and a mobile application (ARCA App).

DETAILED DESCRIPTION:
Primary Objectives:

1. To evaluate the asthma control in children and adolescents with persistent asthma, and its relationship with patient characteristics, treatment and health-related variables (treatment adherence, inhalation technique, inhaler device, asthma triggers, and smoking exposure, among others).
2. To assess the health-related quality of life of children and adolescents with persistent asthma, and its relationship with patient characteristics, treatment and health-related variables (asthma control, treatment adherence and inhalation technique, inhaler device, asthma triggers, and smoking exposure, among others).
3. To assess the risk of severe asthma exacerbations in children and adolescents with persistent asthma and its relationship with patient characteristics, treatment, and health-related variables (asthma control, treatment adherence and inhalation technique, inhaler device, health-related quality of life, asthma triggers, and smoking exposure, among others).

Secondary Objectives:

1. To evaluate the effect of monitoring inhalation techniques on patients' performance according to recommended actions when using inhalers, and outcomes such as asthma control, health-related quality of life, and asthma exacerbations.
2. To assess the treatment adherence in children and adolescents with persistent asthma, and its relationship with other treatment-related factors (inhaler technique, inhaler device, adherence attitudes, and beliefs about illness, inhaler and exacerbations, among others).
3. To evaluate health inequalities in children and adolescents with asthma in Spain.

ARCA is a prospective multicenter observational study in children and adolescents with a clinical diagnosis of persistent asthma. This clinical diagnosis of asthma is defined as the presence of wheezing three times in the last year that improves with the use of bronchodilators. Participants are consecutively recruited in outpatient pediatric pulmonology hospital consultations and primary care physicians.

Patient-reported information is obtained by computer-assisted telephone interviews (CATI) and a mobile application (ARCA App). Telephone interviews are performed by trained interviewers to children 8-16 years old and parents/caregivers of children 6-7 years of age, immediately after recruitment and every 6 months. It includes the evaluation of asthma control, prescribed asthma treatment, adherence, and severe asthma exacerbations. Information about inhalation techniques, socioeconomic status, smoking exposure, triggers, use of peak flow, symptom diary, perceived asthma care, adherence attitudes, and beliefs about illness, inhaler and exacerbations is also collected.

The 'ARCA app' combines 3 age versions: parents/guardians (proxy response) for children 6-7 years old, children aged 8-11 years (self-response), and adolescents aged 12-16 years (self-response). The application consists in an interactive chat, simulating a conversation by Short Message Service (SMS) or Instant Messaging Application (WhatsApp) with someone in real time. It includes the monthly administration of 2 questions (global rating of change and severe asthma exacerbations). At the beginning, after downloading the app, and every two months different standardized questionnaires are administered by turns: the EuroQol (EQ-5D), the Pediatric Asthma Impact Scale (PAIS), inhalation techniques scale, and environment support. These latter scales are administered randomly to two groups of equal size, defined within the subsample recruited by each pediatrician.

All the information that each participant answers through the app can be viewed by the pediatrician through a specific platform. The results of the different questionnaires are shown in charts reflecting the patient's answers over time, using the traffic lights code: green for good outcomes, amber for intermediate, and red for poor. Clinical data is registered at recruitment and annually during the follow-up.

Sample size: To detect differences between two groups in the Asthma Control Questionnaire score of 0.3 SD, 175 patients per group would be required to have a statistical power of 80%, at a significance level of 5%.

ELIGIBILITY:
Inclusion Criteria:

* Children or adolescents aged 6-14.
* Clinical diagnosis of asthma.
* Undergoing treatment with inhaled corticosteroids (alone or combined with long-acting beta-agonists) for more than 6 months in the previous year.
* With access to a smart phone (their own, or their parents').

Exclusion Criteria:

* Concomitant respiratory diseases:
* Chronic obstructive pulmonary disease
* Cystic fibrosis
* Pulmonary fibrosis
* Bronchiectasis
* Active tuberculosis,
* Immunodeficiency associated with alpha 1 antitrypsin deficiency
* Ciliary diseases

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Spanish children and adolescents with persistent asthma seen in the outpatient pediatric pulmonology clinics and primary care pediatricians.
Sampling Method: Non-Probability Sample
Enrollment: 525 (Estimated)
Dates: Start 2017-07-26 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in symptoms control, measured with the Asthma Control Questionnaire (ACQ) | 2, 5, 7 and 10 years after inclusion
  Symptoms control is measured with the Asthma Control Questionnaire (ACQ-symptoms) only, which assesses the frequency of 5 asthma symptoms (night-time waking, symptoms on waking, activity limitation, shortness of breath, and wheeze) during the previous week on a 7-point Likert scale from 0 (no impairment) to 6 (maximum impairment). The overall score, calculated as the mean of item responses, ranges from 0 to 6. A score >1.5 is considered not well-controlled asthma, and scores <0.75 well-controlled asthma.
Change from baseline in Health-Related Quality of Life, measured with the EuroQol | 2, 5, 7 and 10 years after downloading the ARCA app
  The EQ-5D consists of 5 dimensions ("mobility", "looking after myself", "doing usual activities", "having pain/discomfort" and "feeling worried/sad/unhappy). It includes also a visual analogue scale (EQ-VAS) on the general health status from 0 (worst health status) to 100 (best health status possible). The EQ-5D index ranges from 1 (best health state) to negative values (health states valued as worse than death), where 0 is equal to death, allowing the calculation of Quality-Adjusted Life-Years (QALYs).
Number of severe asthmatic exacerbations | 5 and 10 years after inclusion
  As a screening to detect asthma exacerbation, the experience of asthma worsening question is administered through the ARCA app: "In the last month, have you had to take any pill, syrup, oral solution or go to the doctor or hospital, due to asthma worsening?" (Yes/No). If the answer is "yes", a phone call confirms or discards a severe asthma exacerbation through the following questions: "Did you visit or phone your general practitioner, out-of-hours, or walk-in center because your asthma got worse?", "Did you call an ambulance or go to the hospital because of your asthma?", "Did you take steroids tablets (such as Prednisolone or Deltacortril) for at least 2 days because of your asthma?" If the participant answers "yes" to at least one of the 3 questions, an asthma exacerbation is confirmed. These questions were constructed applying the definition of the American Thoracic Society and the European Respiratory Society.

SECONDARY OUTCOMES:
Change from baseline in adherence to the treatment, measured with the Medication Intake Survey adherence scale-Asthma (MIS-A) | 2, 5, 7 and 10 years after inclusion
  Adherence is assessed separately for each controller inhaler, based on self-reported prescription start date, daily dosage recommendations and 3 questions on controller use over increasing time periods (day before, previous week, and previous month). Percentages of medication used versus prescribed are calculated first for each question, and subsequently as composite scores (0-100). The total score is categorized into complete (100%), intermediate, and low (50%) adherence. Medication abuse (temporary occasional) is also evaluated for each treatment.
Change from baseline in quality of the inhaler technique, measured with the Inhalation Technique Scale | 2, 5, 7 and 10 years after downloading the ARCA app
  The Inhalation Technique Scale includes five questions on how often participants perform recommended actions when using inhalers, on a 5-point Likert scale from 0 (never) to 4 (always). The overall score, calculated as the mean of items responses, ranges from 0 to 4 points. Higher values indicate better inhaler technique.
Change from baseline in the Pediatric Asthma Impact Scale (PAIS) | 2, 5, 7 and 10 years after downloading the ARCA app
  The Patient-Reported Outcomes Measurement Information System (PROMIS) developed the short version of the Pediatric Asthma Impact Scale (PAIS), composed of 8 items assessing the past seven days in a 5-point response scale with the options: never, almost never, sometimes, often, and almost always. The total raw score (adding the values of the response to each question) is translated into a T-score with a mean of 50 and a standard deviation (SD) of 10. A score lower than 50 is one SD lower than the mean of the reference population.

CONTACTS AND LOCATIONS:
Overall Officials: Montse Ferrer Fores, MD,PhD, Principal Investigator — Parc de Salut Mar
Locations (15):
- Spain (15):
  - Centro de Salud de Jerez Sur, Cadiz, Andalusia
  - Centro de Salud La Candelaria, Seville, Andalusia
  - Centro de Salud Torre Ramona, Zaragoza, Aragon
  - Hospital Miguel Servet, Zaragoza, Aragon
  - Hospital Universitario Araba, Alava, Basque Country
  - Centro de Salud Dobra, Torrelavega, Cantabria
  - Health Services Research Group, IMIM-Hospital del Mar Medical Research Institute, Barcelona, Catalonia
  - Hospital del Mar, Barcelona, Catalonia
  - Centro de Atención Primaria de la Vila Olímpica, Barcelona, Catalonia
  - Hospital Vall d'Hebron, Barcelona, Catalonia
  - Hospital Parc Taulí, Barcelona, Catalonia
  - Centro de Salud Segovia, Madrid, Madrid
  - Centro de Salud Canillejas, Madrid, Madrid
  - Centro de Salud Dos de Mayo Móstoles, Madrid, Madrid
  - Centro de Salud República de Argentina, Valencia, Valencia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Recruitment platform — http://arca.imim.es